CLINICAL TRIAL: NCT04568499
Title: Presenting Nutrition Characteristics, Comorbidities and Outcomes of COVID-19 in African Humanitarian Settings: a Prospective Cohort Study in South Sudan and DRC
Brief Title: Presenting Nutrition Characteristics, Comorbidities and Outcomes of COVID-19 in African Humanitarian Settings
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Medical Corps (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 13736
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: COVID-19 risk factors; COVID-19 outcomes; Africa; South Sudan; Democratic Republic of the Congo; Humanitarian
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected and Confirmed COVID-19 cases: Suspected and confirmed COVID-19 cases (age 5 years and above) identified at health facilities or via mobile teams in Juba, South Sudan and in Eastern Democratic Republic of the Congo.

SUMMARY:
This study will characterize risk factors for poor COVID-19 outcomes (hospitalization, death) and clinical progression of hospitalized COVID-19 patients in South Sudan and Eastern Democratic Republic of the Congo.

DETAILED DESCRIPTION:
A prospective cohort design will be used to follow suspected, probable, and confirmed COVID-19 cases presenting for care at International Medical Corp [supported] health facilities in Juba, South Sudan and the Kivus in Eastern Democratic Republic of the Congo (DRC). This research seeks to assess risk factors for poor outcomes and characterize clinical disease progression of COVID-19 cases in resource-poor humanitarian contexts in Africa. Specifically, this study aims to characterize risk factors for poor COVID-19 outcomes, including both co-morbidities with evidence from high income settings, as well as prevalent conditions in humanitarian settings (e.g., acute malnutrition, malaria, HIV) for which data is not yet available. This research also aims to determine how the progression of confirmed COVID-19 cases in resource-poor African settings may differ from other settings where data are available.

ELIGIBILITY:
Inclusion Criteria:

* Suspected, probable, and confirmed COVID-19 cases presenting for care at participating health facilities (either by walk-in, referral or transfer) or identified by mobile contact tracing teams.

Exclusion Criteria:

* Individuals unable or unwilling to give informed consent (e.g., due to mental impairment)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children >=5 years of age residing in catchment areas of participating health facilities and mobile contact tracing teams in Juba, South Sudan and in Eastern Democratic Republic of the Congo.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Hospitalization | patients will be followed until asymptomatic or deceased (an average of approximately 1 month)
  Hospitalization due to COVID-19 (proportion of participants hospitalized and risk factors for hospitalization)
Mortality | patients will be followed until asymptomatic or deceased (an average of approximately 1 month)
  Death due to COVID-19 (proportion of participants deceased and risk factors for death)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Doocy, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- Democratic Republic of the Congo (2):
  - Goma General Hospital, Goma
  - Bukavu General Hospital, Kinshasa
- Dr John Garang Infectious Diseases Unit, Juba, South Sudan

IPD SHARING:
Plan to Share IPD: Yes
A limited de-identified data set will be posted on humanitarian data exchange.
Time Frame: Upon completion of analysis and publication of the results, the data will be made publicly available.
Access Criteria: None - data will be accessible via Humanitarian Data Exchange
URL: https://data.humdata.org/

REFERENCES:
- [Derived] Leidman E, Doocy S, Heymsfield G, Sebushishe A, Mbong EN, Majer J; IMC-CDC COVID-19 Research Team; Bollemeijer I. Risk factors for hospitalisation and death from COVID-19: a prospective cohort study in South Sudan and Eastern Democratic Republic of the Congo. BMJ Open. 2022 May 18;12(5):e060639. doi: 10.1136/bmjopen-2021-060639. PMID 35584876